CLINICAL TRIAL: NCT06595459
Title: A Randomized Comparative Effectiveness Trial of Nicotine Pouches for Cigarette Substitution: A Question of Public Health
Brief Title: The Options 2 Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1016; A534253 (Other: UW Madison); Protocol Version 8/22/25 (Other: UW Madison); 1R01CA291761-01 (NIH)
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-07

CONDITIONS: Smoker; Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 3mg Nicotine Pouches (Experimental): Participants will use 3mg nicotine pouches
  Interventions: Drug: Nicotine Pouches
- 6mg Nicotine Pouches (Experimental): Participants will use 6mg nicotine pouches
  Interventions: Drug: Nicotine Pouches
- Nicotine Mini Lozenges (Experimental): Participants will use mini lozenges with dosing based on time to first cigarette (2mg - 4mg)
  Interventions: Drug: Mini Nicotine lozenges
- No Study Product (No Intervention): Participants randomized to this arm will use a mint candy during two different 30-minute laboratory sessions only.

INTERVENTIONS:
Drug: Nicotine Pouches — 3mg or 6mg nicotine pouches
  Other Names: ZYN
  Arms: 3mg Nicotine Pouches; 6mg Nicotine Pouches
Drug: Mini Nicotine lozenges — 2mg to 4mg mini lozenges
  Arms: Nicotine Mini Lozenges

SUMMARY:
The goal of this clinical trial is to investigate how well nicotine pouches and nicotine mini lozenges serve as substitutes for cigarettes when people try to switch from smoking to using these alternate nicotine products.

Participants will:

* Use nicotine pouches, nicotine mini lozenges, or no study product for a week and then try not to smoke for 3 weeks.
* Have 6 in-person research visits and 1 follow-up call
* Complete questionnaires at each study contact and use a smartphone app to record smoking and study product use

DETAILED DESCRIPTION:
Researchers currently lack critical data needed to appraise the potential for nicotine pouches to benefit public health. Specifically, they do not know how readily smokers will adopt pouches, how effectively they can substitute for cigarettes when smokers are trying to avoid smoking, the role of nicotine dose in the ability of pouches to serve as a substitute, or the mechanisms that facilitate or hinder successful product transition. This study will address these questions using a 4-arm randomized controlled trial of adults who smoke ≥5 cigarettes daily and are not planning to quit smoking in the next 30 days. This study will provide a rigorous evaluation of the potential efficacy of a relatively modified risk new nicotine product as a substitute for combusted cigarettes. The head-to-head comparison with FDA-approved mini lozenges can inform tobacco regulatory policy decisions.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 21 years old (i.e., able to legally purchase tobacco products)
* able to read and communicate in English
* no plans to quit smoking in the next 30 days
* willing to stop using nicotine replacement or varenicline
* willing to stop using bupropion (i.e., Wellbutrin, Zyban) if they are currently using it only for smoking cessation
* smoking ≥ 5 cigarettes per day for the past 6 months
* exhaled carbon monoxide ≥ 6 ppm
* no nicotine pouch or smokeless tobacco (including snus) use within the last 6 months

Exclusion Criteria:

* currently in treatment for psychosis or bipolar disorder
* currently taking bupropion for non-smoking cessation reasons (e.g., Wellbutrin for depression)
* currently pregnant or breastfeeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Mean number of cigarettes smoked per day during the 21-day switching period. | Baseline to 3 weeks
  Participants will self-report on their cigarette use

SECONDARY OUTCOMES:
Change in cigarette craving | Baseline to 3 weeks
  Participants will rate their craving for a cigarette using a 0-100 visual analog scale, where 0 = no craving and 100 = extreme craving after sampling their assigned study product after overnight abstinence from smoking
Mean units of study product used per day during the 7-days prior to the switching period | For 7-days leading up to the switching period
  Participants will report their study product use via EMA
Mean units of study product used per day during the 21-day of the switching period | 21-days of the switching period
  Participants will report their study product use via EMA

CONTACTS AND LOCATIONS:
Overall Officials: Megan Piper, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No